CLINICAL TRIAL: NCT00119977
Title: Periacetabular Osteotomy. A Prospective Study With Reference to Cartilage, Migration and Bone Density
Brief Title: Periacetabular Osteotomy.A Prospective Study With Reference to Cartilage, Migration and Bone Density
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Inger Mechlenburg, post doc., Aarhus University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050605
Record Dates: First submitted 2005-07-05; First posted 2005-07-14 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Osteoarthritis
Keywords: cartilage thickness; RSA; DEXA; ultra sound; MRI; osteoarthritis; periacetabular osteotomy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Procedure: 1 Periacetabular osteotomy

INTERVENTIONS:
Procedure: 1 Periacetabular osteotomy — pelvic osteotomy to increase acetabular coverage
  Other Names: periacetabular osteotomy

SUMMARY:
The purpose of this study is to evaluate the effect of performing a periacetabular osteotomy on patients with hip dysplasia.

DETAILED DESCRIPTION:
The cause of osteoarthritis in hip dysplasia is thought to be attributable to increased joint contact pressures secondary to decreased acetabular coverage of the femoral head and/or incongruity of the articular surfaces. The investigators' hypothesis is that when periacetabular osteotomy is performed and contact pressure on cartilage reduced, additional joint degeneration will be slowed or prevented unless irreparable damage to the cartilage has happened at the time periacetabular osteotomy is performed. Hence, the purposes of this study are:

* to develop an unbiased and precise method for measurement of the thickness of the articular cartilage in the hip joint because such a method can be used to evaluate the effect of periacetabular osteotomy and also to give a more precise indication/contraindication for surgery;
* to evaluate the migration of the acetabulum postoperatively and 6 months after surgery by use of RSA to examine the stability of the osteotomy; and
* to examine bone mineral density in acetabulum 1 and 2 years after surgery in order to find out whether the change in load distribution will affect bone density of the acetabulum over time in a way that in the area where more load is applied, bone density will increase, and in areas with less load, bone density will decrease;
* to examine the labrum in the hip joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologically diagnosed hip dysplasia (CE-angle < 25°)
* Patients with osteoarthritis graded 0, 1 or 2 defined according to Tönnis' classification
* Patients with pain from hip
* Age > 18 years
* Minimum 110° flexion in hip joint and closed growth zones in the pelvic region
* Informed consent

Exclusion Criteria:

* Patients with neurological diseases
* Patients with calvé-Legg-Perthes syndrome
* Patients where a femoral intertrochanteric osteotomy is necessary
* Patients with medical sequelae after earlier hip surgery
* Females who are pregnant
* Patients with metal implants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2003-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
migration of acetabulum | six months

SECONDARY OUTCOMES:
BMD in acetabulum | within two and a half year
status of labrum | three years after pelvic osteotomy
changes in cartilage thickness | two and half a year

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD Professor, Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Aarhus Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark